CLINICAL TRIAL: NCT00733434
Title: Phase 4 Study of Postoperative Prostaglandin E1 in Head and Neck Microsurgery
Brief Title: The Use of Prostaglandin E1 in Head and Neck Microsurgery
Acronym: PGE1HNM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yueh-Bih Tang, Professor of Surgery, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200707036R
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Microsurgery; Head and Neck; Prostaglandin E1; Thrombosis; Complications
Keywords: Microsurgery; Head and neck; Prostaglandin E1; Thrombosis; Complication
MeSH Terms: conditions — Thrombosis | interventions — Alprostadil; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients receiving PGE 1 80mcg/500 ml saline continuous intravenous infusion per day after head and neck microsurgery for 5 days
  Interventions: Drug: Prostaglandin E1
- 2 (Placebo Comparator): Patients receiving 500 ml saline continuous intravenous infusion per day after head and neck microsurgery for 5 days
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Prostaglandin E1 — PGE 1 80mcg/500 ml saline continuous intravenous infusion per day after head and neck microsurgery for 5 days
  Other Names: Alprostadil, Promostan
  Arms: 1
Other: Saline — 500 ml saline continuous intravenous infusion per day after head and neck microsurgery for 5 days
  Other Names: Normal saline
  Arms: 2

SUMMARY:
Prostaglandin E1 (PGE1 )has been shown to have vasodilatation and anti-thrombosis effects, so it is used by some surgeons after microsurgery to keep the patency of the anastomosed small vessels. However, PGE 1 may also causes some complications, like pleural effusion or deep vein thrombosis. Therefore, it remains uncertain whether a routine use of PGE 1 after head and neck microsurgery is justified. We aim to test the hypothesis that PGE 1 increases postoperative vessel patency rate in patients undergoing head and neck microsurgery, with a comparable complication rate as the control group.

DETAILED DESCRIPTION:
Despite meticulous microsurgical techniques, free flap failure due to postoperative vessel thrombosis cannot be completely eliminated. Postoperative pharmacological augmentation of the established blood flow is considered as a feasible solution to this problem. Prostaglandin E1 (PGE1 )has been shown to have vasodilatation and anti-thrombosis effects, so it is used by some surgeons after microsurgery to keep the patency of the anastomosed small vessels. However, PGE 1 may also causes some complications, like pleural effusion or deep vein thrombosis. Therefore, it remains uncertain whether a routine use of PGE 1 in every patient after head and neck microsurgery is justified. We aim to test the hypothesis that PGE 1 increases postoperative vessel patency rate in patients undergoing head and neck microsurgery, and yielded a comparable complication rate as the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring microvascular reconstruction after head and neck cancer resection

Exclusion Criteria:

* Patients with coagulation dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Free flap re-exploration rate | 7 days after microsurgery

SECONDARY OUTCOMES:
Surgical complication rate | hospitalization period

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Bih Tang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Disa JJ, Polvora VP, Pusic AL, Singh B, Cordeiro PG. Dextran-related complications in head and neck microsurgery: do the benefits outweigh the risks? A prospective randomized analysis. Plast Reconstr Surg. 2003 Nov;112(6):1534-9. doi: 10.1097/01.PRS.0000083378.58757.54. PMID 14578781
- [Background] Rodriguez Vegas JM, Ruiz Alonso ME, Teran Saavedra PP. PGE-1 in replantation and free tissue transfer: early preliminary experience. Microsurgery. 2007;27(5):395-7. doi: 10.1002/micr.20377. PMID 17596843
- [Background] Ashjian P, Chen CM, Pusic A, Disa JJ, Cordeiro PG, Mehrara BJ. The effect of postoperative anticoagulation on microvascular thrombosis. Ann Plast Surg. 2007 Jul;59(1):36-9; discussion 39-40. doi: 10.1097/01.sap.0000264837.15110.2f. PMID 17589257
- [Background] Watanabe H, Anayama S, Horiuchi T, Sato E, Hamada Y, Ishihara H. Pleural effusion caused by prostaglandin E1 preparation. Chest. 2003 Mar;123(3):952-3. doi: 10.1378/chest.123.3.952. PMID 12628901
- [Background] Barthelmes L, Chezhian C, Aihaku EK. Deep venous thrombosis and venous thrombophlebitis associated with alprostadil treatment for erectile dysfunction. Int J Impot Res. 2002 Jun;14(3):199-200. doi: 10.1038/sj.ijir.3900853. PMID 12058249
- [Background] Lee KS, Suh JD, Han SB, Yoo JC, Lee SJ, Cho SJ. The effect of aspirin and prostaglandin E(1) on the patency of microvascular anastomosis in the rats. Hand Surg. 2001 Dec;6(2):177-85. doi: 10.1142/s0218810401000643. PMID 11901464